CLINICAL TRIAL: NCT02998697
Title: The Effect of Short Term Oral Iron Supplementation in Systolic Heart Failure Patients Suffering From Iron Deficiency Anemia
Brief Title: Short Term Oral Iron Supplementation in Systolic Heart Failure Patients Suffering From Iron Deficiency Anemia
Acronym: IRON5
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Lita Dwi Suryani, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/077/KEP.033EV
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Heart Failure, Systolic; Iron-deficiency Anemia
Keywords: Systolic Heart Failure; Anemia; Iron Deficiency
MeSH Terms: conditions — Heart Failure, Systolic; Anemia, Iron-Deficiency; Anemia; Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated Group (Experimental): Systolic heart failure patients received Ferrous Sulfate 200 mg t.i.d for 90 days
  Interventions: Drug: Ferrous Sulfate
- Control Group (Placebo Comparator): Systolic heart failure patients received placebo oral capsule t.i.d for 90 days
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Ferrous Sulfate — Ferrous sulfate 200 mg t.i.d for 90 days
  Other Names: Ferrous Sulfate oral capsule
  Arms: Treated Group
Drug: Placebo Oral Capsule — Lactose 200 mg t.i.d for 90 days
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine the efficacy of Ferrous Sulphate (FS) tablets in improving iron stores and functional capacity in HF patients with Iron Deficiency Anemia (IDA).

DETAILED DESCRIPTION:
The investigators conducted a double blind randomized controlled trial (RCT) enrolling 54 Heart Failure (HF) patients (LVEF < 50%) with IDA (Ferritin < 100 ng/mL or 100-300 ng/mL with Tsat < 20%) at outpatient clinic of National Cardiovascular Center Harapan Kita from January to July 2016. Patients were randomized 1:1 to received FS or placebo for 90 days, the investigators then evaluated the change in 6-Minute Walking Test (6MWT) distance as primary end-point and changes on N-Terminal-pro Brain Natriuretic Peptide (NT-proBNP) and post 6MWT serum lactate levels as secondary end-points.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year old
* Systolic heart failure patients without clinical sign of decompensation at outpatient clinic
* New York Heart Association (NYHA) functional class II-III able to perform 6MWT
* LVEF < 50%
* On heart failure therapy
* Haemoglobin (Hb) < 13 gr/dL (male); Hb < 12 gr/dL (female) and > 8 gr/dL
* Ferritin < 100 µg/L or Ferritin 100-300 µg/L dengan Transferrin saturation (Tsat) < 20%
* Agree to participate

Exclusion Criteria:

* History of : active bleeding,infection, malignancy, haematological abnormality, peptic ulcer
* History of myocardial revascularization (CABG/PCI) within 3 month
* Acute Coronary Syndrome (ACS), stroke,Transient Ischemic Attack (TIA) within 3 month
* Know to have allergic reaction to Ferrous sulfate
* History of intravenous iron administration within 1 month
* Permanent Pace Maker(PPM)/Implantable Cardiac Defibrillator (ICD)/Cardiac Resynchronization Therapy (CRT)
* estimated Glomerular Filtration Rate (eGFR) < 30 ml/min/1.73m2
* NT-proBNP > 4000 pg/ml (for patients without baseline data) or decreased level of NT-proBNP < 30% from baseline
* Increase level of serum alanine aminotransferase (ALT)/ serum aspartate aminotransferase (AST)> 3x normal value
* Moderate to severe primary valvular heart disease
* Congenital heart disease
* Right heart failure due to primary pulmonary hypertension, cor pulmonale, Chronic Thrombo-Embolic Pulmonary Hypertension (CTEPH)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 90 days
  Six Minute Walk Test (meter)

SECONDARY OUTCOMES:
Ferritin | 90 days
  Ferritin level (ng/mL)
Transferrin saturation | 90 days
  Transferrin saturation (%)
Haemoglobin | 90 days
  Haemoglobin level (gr/dL)
Echocardiography parameters | 90 days
  Left Ventricle Ejection Fraction
N Terminal-pro Brain Natriuretic Peptide | 90 days
  NT-proBNP level (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Bambang B Siswanto, Professor, Study Director — National Cardiovascular Center Harapan Kita

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Niehaus ED, Malhotra R, Cocca-Spofford D, Semigran M, Lewis GD. Repletion of Iron Stores With the Use of Oral Iron Supplementation in Patients With Systolic Heart Failure. J Card Fail. 2015 Aug;21(8):694-7. doi: 10.1016/j.cardfail.2015.05.006. Epub 2015 May 29. PMID 26028263
- [Result] Anker SD, Comin Colet J, Filippatos G, Willenheimer R, Dickstein K, Drexler H, Luscher TF, Bart B, Banasiak W, Niegowska J, Kirwan BA, Mori C, von Eisenhart Rothe B, Pocock SJ, Poole-Wilson PA, Ponikowski P; FAIR-HF Trial Investigators. Ferric carboxymaltose in patients with heart failure and iron deficiency. N Engl J Med. 2009 Dec 17;361(25):2436-48. doi: 10.1056/NEJMoa0908355. Epub 2009 Nov 17. PMID 19920054
- [Result] McDonagh T, Macdougall IC. Iron therapy for the treatment of iron deficiency in chronic heart failure: intravenous or oral? Eur J Heart Fail. 2015 Mar;17(3):248-62. doi: 10.1002/ejhf.236. Epub 2015 Jan 30. PMID 25639592
- [Derived] Suryani LD, Raharjo SB, Sagita R, Angkasa H, Prasetyadi YL, Suyatna FD, Hersunarti N, Soerarso R, Siswanto BB, Muliawan HS. Oral Ferrous Sulphate Improves Functional Capacity on Heart Failure Patients with Iron Deficiency Anemia. Glob Heart. 2022 Nov 22;17(1):81. doi: 10.5334/gh.1151. eCollection 2022. PMID 36578916